CLINICAL TRIAL: NCT01993485
Title: The Effect of Transaortic Valve Replacement on the Endothelial Integrity and Function
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Other Study IDs: MP TAVI
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Degenerative Aortic Valve Stenosis
Keywords: transaortic valve replacement (TAVI); endothelial function; circulating microparticles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Degenerative aortic valve stenosis (AVS) is the leading cause of aortic valve morbidity with a prevalence of 2-7% at ages above 65 years, with ever-increasing incidence especially in the 8th decades. AVS is independently associated with atheroclerosis risk factors and clinically apparent CV disease indicating that the degeneration of the aortic valve may represent an atheroclerosis-like process involving both, the aortic valve as well as the vascular system, respectivel. It is still unknown whether the endothelial function is affected as an manifestation of the atherosclerotic process, changes in the driving mechanical forces as WSS downstream of the valve, or other factors beyond physical pressure effects.

The investigators hypothesized that altered haemodynamics may at least partly be responsible for observed endothelial dysfunction in patients with AVS. Therefore, the aim of this study is to investigate whether the resolution of AVS by transaortic valve implacement (TAVI) affects WSS, improves endothelial dysfunction and decreases levels of circulating EMPs as markers of endothelial integrity.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve stenosis
* screened for TAVI
* written informed consent

Exclusion Criteria:

* no written informed consent
* Patients with acute infections (CRP> 0.5 mg / dL)
* Patients with Atrial Fibrillation
* Patients with inflammatory and malignant diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with aortic valve stenosis screened for TAVI
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
endothelial function | Changes from Baseline in endothelial function at 3 months
  endothelial function will be measured by flow mediated dilation (FMD)
plasma levels of circulating microparticles (MPs) | Changes from Baseline in Plasma Levels of MPs at 3 months

SECONDARY OUTCOMES:
arterial stiffness | Changes from Baseline in arterial stiffness at 3 months
  arterial stiffness will be measured by pulse wave analysis
blood pressure | Changes from Baseline in Hemodynamics at 3 months
heart rate | Changes from Baseline in Hemodynamics at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Westenfeld, MD, Principal Investigator — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Dusseldorf; Malte Kelm, Professor, Study Chair — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Dusseldorf
Locations (1):
- Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Dusseldorf, Düsseldorf, Germany